CLINICAL TRIAL: NCT01311583
Title: Evaluating Teach Back as a Method for Improving Self-Care Behaviours in Heart Failure Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 11-010
Record Dates: First submitted 2011-02-22; First posted 2011-03-09 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Heart Failure
Keywords: Self-care; Teach Back
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- usual care plus Teach Back intervention (Active Comparator): Trained nurses will provide Teach Back to the intervention group. The nurses' training will focus on the concepts of Teach Back, provide coaching and guidance on how to use it as well as review the principles of conducting research. Role play will be a feature in the education sessions to improve the nurses' comfort level
  Interventions: Behavioral: Teach Back method of patient discharge teaching
- usual care (No Intervention): All participants will experience the current practice of discharge teaching: daily interaction with the interdisciplinary team members via rounds, counseling on diet and medications with a dietician and pharmacist when referred, view the Heart Failure Discharge Video, and receive a Congestive Heart Failure education package which includes the Heart and Stroke "Managing Congestive Heart Failure" booklet.

INTERVENTIONS:
Behavioral: Teach Back method of patient discharge teaching — Trained nurses will provide Teach Back to the intervention group. Appendix D lists the four questions that will be used in this study to confirm the patient's understanding. The nurses' training will focus on the concepts of Teach Back, provide coaching and guidance on how to use it as well as review the principles of conducting research. Role play will be a feature in the education sessions to improve the nurses' comfort level
  Arms: usual care plus Teach Back intervention

SUMMARY:
Patient education using Teach Back has the potential to increase self-care behaviour in heart failure (HF) patients and reduce adverse clinical outcomes. Teach back is an interactive teaching method that uses plain language, focuses on key points, and asks the patient to verbally recall information just discussed. Questions are asked to confirm patient understanding of the information delivered.

This pilot study will be conducted to evaluate the effectiveness of teach back on self-care (as measured by the European Heart Failure Self-Care Behaviour Scale- EHFScBS) and determine if teach back affects the number of ER visits and re-admissions post discharge. The study will also assess if teach back technique is a feasible, acceptable and sustainable method of discharge teaching for hospitalized HF patients at St Michael's.

DETAILED DESCRIPTION:
Background: Heart Failure (HF) is a common and debilitating disease associated with frequent hospitalizations, decreased quality of life, and requires complex health care regimen. Heart failure management programs promote self-care by teaching patients how to recognize signs and symptoms, how to respond to these symptoms and who to contact for advice. Teaching interventions aimed at self-care have been shown to improve patient outcomes, however, the optimal method of delivering the education is unknown.

Patient education using Teach Back has the potential to increase self-care behaviour in HF patients and reduce adverse clinical outcomes by using plain language, focusing on key points, and asking the patient to verbally recall information just discussed, in an interactive manner. Research has shown Teach Back to be an effective strategy to improve patient comprehension in chronic conditions such as HF and diabetes.

The RNAO Best Practice Guidelines for Self-Management in Chronic Conditions (2010) recommends a nursing communication technique of "Closing the Loop" also known as "Teach Back" to assess patient understanding of information. The level of evidence for this technique is level III (from well designed, non-experimental descriptive studies, such as comparative studies, correlation studies, and case studies). This study will provide additional evidence in a randomized experimental design.

The objectives of this study are to evaluate the effectiveness of Teach Back on self-care (as measured by the European Heart Failure Self-Care Behaviour Scale) and determine if Teach Back affects the number of ER visits and re-admissions post discharge. A secondary objective is to assess if Teach Back technique is a feasible, accepted and sustainable method of discharge teaching for hospitalized HF patients at St. Michael's.

1. Research Question: Does discharge teaching using the Teach Back method from trained nurses improve self-care behaviour in HF patients as measured by the EHFScBS scale as compared to standard care discharge teaching?

   Hypothesis: Patients who receive teach back discharge teaching will have improved self-care (achieve lower scores on EHFScBS).
2. Research Question: Are there fewer ER visits and hospital admissions post discharge in patients who receive instruction with teach back method?

   Hypothesis: Patients who receive discharge teaching with Teach Back will have less ER visits and hospital admissions in the 3 months following hospital discharge.
3. Research Question: What is the feasibility and acceptability of adapting Teach Back as standard practice of discharge teaching for heart failure patients in the in-patient cardiac care units at St. Michael's?

Hypothesis: Teach Back is an accepted and sustainable method of discharge teaching in HF patients in the in-patient cardiac care units at St. Michael's as evidenced by participants' feedback (patient questionnaires and nursing focus groups).

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the in-patient cardiology (7CCS) or Coronary Care Unit (CCU), with documentation of HF as the most responsible diagnosis
* Prescribed a diuretic such as Lasix plus or minus Metolazone
* New or established diagnosis of HF

Exclusion Criteria:

* Cognitive impairment
* Suffer from a co-existing, severe, chronic debilitating disease
* Require hemo or peritoneal dialysis, have planned surgical intervention that will impact the etiology or manifestation of HF symptoms
* Life expectancy of less than three months
* Unable to receive discharge teaching, or are unable to communicate on the telephone
* Already enrolled in a patient education study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2011-10; Primary Completion 2012-10 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
self-care behaviour score | change from baseline in self-care behaviour score at one week.
  mailed questionaire
self-care behaviour score | change from baseline in self-care behaviour score at one month
  mailed questionaire
self-care behaviour score | change from baseline in self-care behaviour score at three months
  mailed questionaire

SECONDARY OUTCOMES:
patient visits to ER or admission to hospital | one week since discharge
  mailed questionaire
patient visits to ER or admission to hospital | at one month since discharge
  questionaire
patient ER visits or admission to hospital | three months since discharge
  questionaire
impact on nurses' workload | up to 12 weeks from the last enrolled patient
  focus group
satisfaction with the training for the nurses' to provide teach back | up to 12 weeks from the last enrolled patient
  focus group
nurses' conviction and confidence related to Teach Back | up to 12 weeks from the last enrolled patient
  focus group

CONTACTS AND LOCATIONS:
Overall Officials: Ada Andrade, MN, Principal Investigator — St. Michael's; Vimy Barnard-Roberts, MN, Study Chair — St. Michael's; Haytham Sharar, MN, Study Chair — St. Michael's
Locations (1):
- St. Michael's, Toronto, Ontario, Canada